CLINICAL TRIAL: NCT06338605
Title: Evaluating the Incidence of Pseudo-Acute Kidney Injuries in Patients With Metastatic Breast Cancer on CDK4/6 Inhibitors Trough Cystatin C Analysis
Acronym: CYSTATINcDK4/6
Status: Active, not recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Agnes Jager MD, PhD, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2023-0715
Record Dates: First submitted 2024-03-08; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention, observational study of AKI under CDK4/6 inhibitor treatment — no intervention

SUMMARY:
CDK4/6 inhibitors have led to an improvement of both progression free survival (PFS) and overall survival (OS) in patients with advanced estrogen positive (ER+)/HER2- breast cancer when applied in the first or second line of treatment. Despite the advantages of CDK4/6 inhibitors, these medications can lead to adverse effects. One of the adverse events observed across all types of CDK4/6 inhibitors is an elevation in creatinine levels. An elevation in plasma creatinine during treatment with abemaciclib is not always indicative of a reduction in renal function; it can also be attributed to the inhibition of active tubular secretion of creatinine. This phenomenon is known as pseudo acute kidney injury (pseudo-AKI).

The incidence of pseudo-AKI in patients using CDK4/6 inhibitors is currently unknown. A method to distinguish pseudo-AKI from AKI is measuring the level of an alternative filtration marker in blood, for example cystatin C. Cystatin C is also filtered at the glomerulus but not secreted intro the renal tubulus or reabsorbed into the bloodstream. Also, there is no affection by muscle mass or diet. In this study the investigators will explore the incidence of both AKI and pseudo-AKI in patients who are treated with CDK4/6 inhibitor treatment by assessing both creatinine and cystatin C in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are receiving CDK4/6 inhibitors for metastatic breast cancer
* Patients must have used the CDK4/6 inhibitor for a minimum duration of one month
* Patients must have undergone at least one measurement of creatinine after the initiation of CDK4/6 inhibitor treatment

Exclusion Criteria:

- Patients who are undergoing dialysis therapy for kidney failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic breast cancer that are treated with a CDK4/6 inhibitor (i.e. palbociclib, ribociclib, abemaciclib).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pseudo-AKI in patients on CDK4/6 inhibitors | jan-april 2024
  Percentage of patients with pseudo-AKI (%), i.e. patients with creatinin plasma levels (mmol/L) indicating AKI, but normal cystatin C levels (mg/mL)

SECONDARY OUTCOMES:
Pseudo-AKI in patients on CDK4/6 inhibitors per drug | jan-april 2024
  The percentage of patients (%) per CDK4/6 inhibitor with creatinin plasma levels indicating AKI
AKI in patients | jan-april 2024
  The percentage of patients (%) on CDK4/6 inhibitors with cystatin C plasma levels indicating AKI
Influencing factors cystatin C levels | jan-april 2024
  The number of patients with influencing factors on cystatin C levels

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided